CLINICAL TRIAL: NCT00478842
Title: Treatment of Gilles de la Tourette Syndrome by Bilateral Stimulation of the Internal Part of the Globus PALLIDUS
Brief Title: Pallidal Stimulation and Gilles de la Tourette Syndrome
Acronym: STIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P051050
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Gilles de la Tourette Syndrome
Keywords: Gilles de la Tourette syndrome; Deep brain stimulation; Globus PALLIDUS
MeSH Terms: conditions — Tourette Syndrome | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Deep brain stimulation
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Deep brain stimulation

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of bilateral pallidal stimulation in patients with a severe form of Gilles de la Tourette syndrome.

DETAILED DESCRIPTION:
It acts of a randomized study, in parallel, double group blind, multi-centric relating to 14 patients.

The interest of this multicentric study, which will be carried out in centers specialized in the field of major cerebral stimulation with for each one a multidisciplinary team, is to carry out a homogeneous protocol which should make it possible to give a clear response in term of effectiveness for this treatment in this pathology.

The evaluation will be:

1. neurological (YGTSS, video scale of the tics);
2. psychiatric, with in particular of the specific psychopathological evaluations centered on mood;
3. neuropsychological, centered on impulsiveness;
4. functional calculus evaluating total operation and the social adaptation;
5. neurophysiological (recording of the neuronal activities).

Calculations of the number of subjects necessary showed, by laying down the principal objective at an improvement of at least 60 % of the score of the YGTSS under treatment, which 14 subjects will make it possible to show a significant difference with the procedure placebo.

Study in Tomography by Emission of Positrons (Mtoe) carried out on 8 of the 14 operated patients having had at least 3 months of stimulation, in comparison on 8 pilot subjects (paired for the sex and the age), should make it possible to determine, at the time of the improvement of the driving symptoms, modifications of cerebral activation induced by the high frequency stimulation of GPI among patients.

The association of this study to the comparison of the improvement of the neurological symptoms with the precise localization of the therapeutic stud of the electrode reformatted on the post-operative TDM (8), carried out for all the patients, should make it possible to specify the anatomy-physiological bases to specify the anatomy-physiological bases of the MGT The duration of the study will be 14 month for each patient, that is to say one 2 months preoperative period intended for inclusion; one 3 months post-operative period without stimulation; one period randomized with stimulation either "one" (3 months), or "off" (3 months), then an open study for all the patients with stimulation "one" for one 6 months duration.

It is envisaged to include 14 patients reached of the MGT (of which 8 will take part in study Mtoe) and 8 subjects controls for study Mtoe is 22 subjects.

An observational follow-up at 30 and 48 months is added.

ELIGIBILITY:
Inclusion Criteria:

* Severe form of GTS
* age 18 to 60 years
* failure of medical treatment (including neuroleptics)

Exclusion Criteria:

* Major depression
* Psychotic symptoms
* Severe personality disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the therapeutic effect of the high frequency bilateral stimulation of GPI in severe forms and invalidating MGT, in a protocol randomized as a double blind man in parallel groups. | during the 44 months
The assumption tested is that of the frank improvement (> 60% on scale YGTSS) of the symptoms of the MGT by the bilateral stimulation of GPI in its former part. | at the end of 44 months

SECONDARY OUTCOMES:
To evaluate time necessary to obtaining the maximum effect and its evolution after this one (maintenance or not of the effect in the course of time) | during the study
To study the effects of the stimulation of GPI in its former part, on the driving tics simple and complex, vocal, the self-mutilations, and the psychopathology of which time, emotions and impulsiveness | during the 44 months
To evaluate the repercussion of this technique on the sociological-professional handicap, operation and the adaptation | during the 44 months
To seek determinants before intervention of the effectiveness of stimulation (determining neurological, psychiatric, neuropsychological, functional) | during the 44 months
To establish correlations between the localization of the studs of stimulation (retiming atlas/IRM) and the symptoms | during the 44 months
To determine the modifications of cerebral activation induced by the bilateral stimulation of GPI at the time of the improvement of the neurological symptoms (study in Mtoe). | during the 44 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure WELTER, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe hospitalier la Pitié Salpétrière, Paris, France

REFERENCES:
- [Result] Houeto JL, Karachi C, Mallet L, Pillon B, Yelnik J, Mesnage V, Welter ML, Navarro S, Pelissolo A, Damier P, Pidoux B, Dormont D, Cornu P, Agid Y. Tourette's syndrome and deep brain stimulation. J Neurol Neurosurg Psychiatry. 2005 Jul;76(7):992-5. doi: 10.1136/jnnp.2004.043273. PMID 15965209
- [Derived] Welter ML, Houeto JL, Thobois S, Bataille B, Guenot M, Worbe Y, Hartmann A, Czernecki V, Bardinet E, Yelnik J, du Montcel ST, Agid Y, Vidailhet M, Cornu P, Tanguy A, Ansquer S, Jaafari N, Poulet E, Serra G, Burbaud P, Cuny E, Aouizerate B, Pollak P, Chabardes S, Polosan M, Borg M, Fontaine D, Giordana B, Raoul S, Rouaud T, Sauvaget A, Jalenques I, Karachi C, Mallet L; STIC study group. Anterior pallidal deep brain stimulation for Tourette's syndrome: a randomised, double-blind, controlled trial. Lancet Neurol. 2017 Aug;16(8):610-619. doi: 10.1016/S1474-4422(17)30160-6. Epub 2017 Jun 20. PMID 28645853